CLINICAL TRIAL: NCT02998515
Title: Effects of Supplemental Oxygen Delivery Via Portable Oxygen Concentrator (Activox™4L) vs. Liquid Oxygen Device in Hypoxemic COPD Patients - a Non-inferiority Study
Brief Title: Effects of Different Oxygen Devices in Hypoxemic COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: ResMed (Industry)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician of the department of Pneumology, Schön Klinik Berchtesgadener Land
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ACT2016
Record Dates: First submitted 2016-12-01; First posted 2016-12-20 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Chronic Obstructive Pulmonary Disease Severe
Keywords: supplemental oxygen; concentrator; endurance shuttle walk test

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ESWT order: 1.liquid oxygen, 2. concentrator (Experimental): Patients will start with the endurance shuttle walk test (ESWT) by using supplemental Oxygen from a portable liquid Oxygen device (Companion) and continue on the day after with ESWT by using supplemental Oxygen from a portable concentrator.
  Interventions: Device: Companion (Liquid oxygen device); Device: Activox (concentrator)
- ESWT order: 1. concentrator, 2. liquid oxygen (Experimental): Patients will start with the endurance shuttle walk test (ESWT) by using supplemental Oxygen from a concentrator and continue on the day after with ESWT by using supplemental Oxygen from a portable liquid Oxygen device.
  Interventions: Device: Companion (Liquid oxygen device); Device: Activox (concentrator)

INTERVENTIONS:
Device: Companion (Liquid oxygen device)
  Other Names: Device: Companion
Device: Activox (concentrator)
  Other Names: Device: Activox

SUMMARY:
Taken recent literature together, there is a sufficient number of trials investigating the effect of different oxygen devices. However, studies comparing oxygen delivery via portable oxygen concentrator (POC) and liquid oxygen device (LOD) with appropriate exercise testing and sufficient power are missing.

Given that walking is the most important activity of daily life to preserve the maintenance and to participate in social life, we aim to investigate the effects of two different oxygen delivery systems during walking in hypoxemic COPD patients (POC vs. LOD).

The endurance shuttle walk test (ESWT) is well validated for measuring endurance walking capacity in COPD patients with good repeatability. The advantage of this test over the 6MWT is that the ESWT is performed at 85% of the individual maximum which is close to the intensity of typical daily activities. Due to the fact that the ESWT enables us to determine the maximum duration of exercise and to compare values at isotime (at the point of time when the shortest of the 3 ESWTs ends), we use the ESWT as exercise test in our trial.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients (GOLD stage III to IV) with hypoxemia at rest or during exercise (paO2<60mmHg)
* Participation in an inpatient pulmonary rehabilitation program (Schön Klinik BGL)
* Written informed consent

Exclusion Criteria:

* General exclusion criteria for exercise tests, e.g. acute coronary syndrome, acute myo- or pericarditis, acute lung embolism, pulmonary infarction, acute uncontrolled heart insufficiency
* Signs of acute exacerbation
* Any orthopedic or neurological disabilities that prevent patient from walking

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in oxygen Saturation during endurance shuttle walk test (ESWT) compared between POC (concentrator) and LOD (liquid oxygen) | Change from baseline to the individual end of ESWT (until exhaustion, max. 20 minutes)
  ESWT is designed to assess the Maximum Walking Duration that can be sustained at 85% of individual Maximum capacity. Therefore, outcome Parameter will also be assessed at the individual end of the ESWT.

SECONDARY OUTCOMES:
Change in Breathing frequency | Change from baseline to the individual end of ESWT (until exhaustion, max. 20 minutes)
  ESWT is designed to assess the Maximum Walking Duration that can be sustained at 85% of individual Maximum capacity. Therefore, outcome Parameter will also be assessed at the individual end of the ESWT.
Change in Inspiratory capacity | Change from baseline to the individual end of ESWT(until exhaustion, max. 20 minutes)
  ESWT is designed to assess the Maximum Walking Duration that can be sustained at 85% of individual Maximum capacity. Therefore, outcome Parameter will also be assessed at the individual end of the ESWT.
  Inspiratory capacity will be measured by a mobile spirometry (SpiroPalm mask).
Endurance shuttle walk distance | at the end of ESWT (until exhaustion, max. 20 minutes)
  ESWT is designed to assess the Maximum Walking Duration that can be sustained at 85% of individual Maximum capacity.
Change in perceived Dyspnea | Change from baseline to the individual end of ESWT (until exhaustion, max. 20 minutes)
  ESWT is designed to assess the Maximum Walking Duration that can be sustained at 85% of individual Maximum capacity. Therefore, outcome Parameter will also be assessed at the individual end of the ESWT. Dyspnea will be rated by the Patient on a 10-point Borg scale.
Change in partial pressure of carbon dioxide | Change from baseline to the individual end of ESWT (until exhaustion, max. 20 minutes)
  ESWT is designed to assess the Maximum Walking Duration that can be sustained at 85% of individual Maximum capacity. Therefore, outcome Parameter will also be assessed at the individual end of the ESWT.

CONTACTS AND LOCATIONS:
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany

IPD SHARING:
Plan to Share IPD: Undecided